CLINICAL TRIAL: NCT05717283
Title: Follow-up of the Nasal Microbiome and Viral Infections in Newborns Hospitalised in Neonatology in the University Hospital of Caen, France : Metatranscriptomics Approach by Next Generation Sequencing From Nasal Swabs.
Brief Title: Follow-up of the Nasal Microbiome and Viral Infections in Newborns Hospitalised in Neonatology.
Acronym: NEOBIOME
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2022-A01965-38
Record Dates: First submitted 2023-01-04; First posted 2023-02-08 (Actual); Last update posted 2024-02-13 (Actual); Status verified 2024-01

CONDITIONS: Microbial Colonization; Viral Infection; Neonatal Infection
Keywords: Metatranscriptomics; Microbiome; Newborn
MeSH Terms: conditions — Communicable Diseases; Virus Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Nasal swab — We will take nasal swabs from anterior and middle nostril, once a week for each newborn included.

SUMMARY:
The goal of this interventional study is to learn about nasal microbiome and viral infections in newborns hospitalised in neonatology.

The main questions it aims to answer are :

* how often are newborns infected by viruses in neonatology ?
* how does the microbiome develop during first weeks of life ?
* how does microbiome and viruses interacts together ?
* is there a link between viral infection, microbiome, and medical complications during hospitalisation in neonatology ? Participants will have a nasal swab taken each week during their hospitalisation in neonatology, and researchers will take medical data from the medical chart.

ELIGIBILITY:
Inclusion Criteria:

* newborn hospitalised in neonatal intensive care unit during the inclusion period
* parents have been informed about the study (speaking french) and have signed the informed consent.
* affiliated to the social security system.

Exclusion Criteria:

* parental refusal
* minor parents or under judicial protection
* newborn who already have been discharded home before inclusion
* hospitalisation after the first 48 hours of life
* only palliative care

Max Age: 48 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 38 (Actual)
Dates: Start 2022-12-20 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
Change in microbiome diversity | Day 0, day 7, day 14, and each week until discharge (maximum duration : 3 months for each newborn).
  Shannon diversity index
Change in microbiome abundance | Day 0, day 7, day 14, and each week until discharge (maximum duration : 3 months for each newborn).
  Number of reads for a given taxonomy.
Virus presence | Day 0, day 7, day 14, and each week until discharge (maximum duration : 3 months for each newborn).
  Molecular detection of respiratory viruses using multiplex PCR.

SECONDARY OUTCOMES:
Occurence of bronchopulmonary dysplasia | At discharge from neonatology.
  assessed by clinical recording on discharge from neonatology
Change in expression of local innate immunity markers | Day 0, day 7, day 14, and each week until discharge (maximum duration : 3 months for each newborn).
  Mesure of the expression of the interferon-stimulated genes (ISGs), anti-viral genes, and the inflammasome pathway.

CONTACTS AND LOCATIONS:
Locations (1):
- CAEN University Hospital, Caen, France

IPD SHARING:
Plan to Share IPD: No
Individual participant data will be anonymised.